CLINICAL TRIAL: NCT04161040
Title: Laboratory Model for Relapse to Sedentary Behavior: Toward a Physically Active West Virginia
Brief Title: Laboratory Model for Relapse to Sedentary Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1810337844
Record Dates: First submitted 2019-11-04; First posted 2019-11-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Exercise
Keywords: Relapse; Physical Activity; Sedentary Behavior; Behavioral Momentum Theory; Incentives
MeSH Terms: conditions — Motor Activity; Recurrence; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Block randomization will be used to assign participants to one of three groups (one experimental and two control groups). All groups will experience three phases of the study. Opportunities for sedentary leisure and physical activities will be continuously available throughout all phases.
Who Masked: Participant
Masking Description: The participants will not be told which group they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relapse (experimental) Group (Experimental): Opportunities for sedentary leisure and physical activities will be continuously available throughout all phases. Each phase will last 20 minutes. The first phase will mimic pre-intervention conditions; there will be a variety of activities available. No incentives for engaging in physical activity will be provided, although such activities will be available. For the Relapse (experimental) Group, the second phase will mimic an incentive-based intervention in which participants can earn monetary incentives for engaging in physical activity. Then, during the third phase, the incentives will be discontinued.
  Interventions: Behavioral: Performance-based incentives
- Fatigue Control Group (Experimental): Opportunities for sedentary leisure and physical activities will be continuously available throughout all phases. Each phase will last 20 minutes. The first phase will mimic pre-intervention conditions; there will be a variety of activities available. No incentives for engaging in physical activity will be provided, although such activities will be available. The second phase will mimic an incentive-based intervention in which participants can earn monetary incentives for engaging in physical activity. Participants in this arm will continue to earn incentives during Phase 3 to control reductions in physical activity due to fatigue.
  Interventions: Behavioral: Performance-based incentives
- No-Incentive Control Group (No Intervention): Opportunities for sedentary leisure and physical activities will be continuously available throughout all phases. Each phase will last 20 minutes. Participants in this arm will not earn incentives during any of the three phases to control for the possibility that participants will engage in some physical activity in the absence of incentives.

INTERVENTIONS:
Behavioral: Performance-based incentives — Participants will earn $1 per minute of engagement in physical activity.
  Arms: Fatigue Control Group; Relapse (experimental) Group

SUMMARY:
Physical inactivity is a key risk factor for noncommunicable illnesses such as cancer and cardiovascular disease-the two leading causes of death in West Virginia. The World Health Organization recommends muscle-strengthening activities 2 or more days per week and a minimum of either 150 minutes of moderate-intensity activity or 75 minutes of vigorous-intensity activity per week. Yet, only one in five adults in the United States meets these recommendations. Even more alarming is that 33.2% of West Virginians report that they did not engage in any physical activity in the past month. Incentive-based interventions increase physical activity in the short term, but incentives for healthy behavior are generally discontinued after some period of time, and relapse of unhealthy behavior is common. Thus, there is a critical need to develop interventions that result in both immediate and lasting engagement in activity. The overall objective and specific aim of the proposed project is to evaluate a brief laboratory model of relapse into sedentary behavior following incentive-based interventions that is based on Behavioral Momentum Theory. The central hypothesis is that incentives will increase activity, but relapse will occur in the brief model, like what occurs in extended clinical treatment. Development of a laboratory model of relapse into sedentary behavior (the expected outcome of the proposed project) will inform future translational research, eventually leading to clinical applications of large-scale physical-activity interventions that result in significant and immediate behavior change and that minimize relapse.

DETAILED DESCRIPTION:
Physical inactivity is a key risk factor for noncommunicable illnesses such as cancer and cardiovascular disease (CVD)-the two leading causes of death in West Virginia. Physical inactivity is fundamentally a behavior problem, and there is a growing body of research supporting the use of incentive-based interventions to increase physical activity. In such interventions, participants earn incentives such as money, tokens or points, entries into prize drawings, or fitness-related commodities (e.g., gym memberships) by meeting defined goals (e.g., daily steps, energy expenditure, fitness classes).

A crucial feature of any successful intervention is sustained behavior-change following the removal or decrease in supports. However, most evaluations of incentive-based interventions are completed on a short-term scale (4 to 12 weeks) and often fail to provide data on follow-up. The studies that follow participants after the discontinuation of incentives often show relapse to sedentary behavior following intervention. Similar relapse is common following incentive-based interventions for other health-related behavior. Laboratory models of relapse prevention have informed treatment for these other forms of health-related behavior, but they have yet to be extended to interventions addressing sedentary behavior.

The investigators' long-term goal is to develop practical interventions that sustain increases in physical activity and thereby decrease a significant risk factor for disease (e.g., cancer, diabetes). The overall objective of the proposed project is to evaluate a brief laboratory model of relapse that is based on basic behavioral research grounded in Behavioral Momentum Theory. The central hypothesis is that incentives in the brief model will produce the expected increases in physical activity relative to no-incentive controls, but that these gains will be rapidly lost when the incentives are discontinued. This hypothesis is based other laboratory-based models of relapse (e.g., illicit drug use and challenging behavior), which mirrored outcomes of, and led to advances in clinical, treatment. The rationale for this project is that a laboratory model of relapse of sedentary behavior will inform future translational research and lead to large-scale clinical trials of incentives to improve physical activity that result in large, immediate behavioral change and that minimize subsequent relapse.

The central hypothesis is that incentives in the brief model will produce the expected increases in physical activity relative to no-incentive controls, but that these gains will be rapidly lost when the incentives are discontinued. These outcomes would suggest that the brief model produces outcomes similar to those obtained in more extended clinical treatment.

Approach The anticipated number of participants is 30 individuals (age 18-74). Participants will attend a single 90-min laboratory appointment. The laboratory space will be equipped with a treadmill, comfortable seating, and leisure activities. A licensed nurse will screen participants to ensure they are healthy enough to engage in physical activity and will remain present for the duration of participation to provide medical assistance in the unlikely event that it is needed. Block randomization will be used to assign participants to one of three groups (one experimental and two control groups). All groups will experience three phases of the study. Opportunities for sedentary leisure and physical activities will be continuously available throughout all phases. The first phase will mimic pre-intervention conditions; there will be a variety of activities available. No incentives for engaging in physical activity will be provided, although such activities will be available. For the Relapse (experimental) Group, the second phase will mimic an incentive-based intervention in which participants can earn monetary incentives for engaging in physical activity. Then, during the third phase, the incentives will be discontinued the Fatigue Control group will experience the same conditions for Phase 1 and 2, but they will continue to earn incentives during Phase 3. The No-Incentive Control group will not earn incentives during any phase to control for the possibility that participants will engage in some physical activity in the absence of incentives.

Participants will wear a heart rate monitor throughout the study to provide real-time data on activity level and trained research assistants will use software to score time-stamped duration of engagement in available activities (e.g., walking, sitting). A one-way ANOVA will be used to compare mean durations of physical activity across groups. A power analysis[23] shows that including 30 participants (10 in each group) will provide sufficient power to detect an effect size of 0.8 at an alpha of 0.05. Additionally, the investigators will use the heart rate data for preliminary analyses of mediation and moderation effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults of any gender between the ages of 18 and 74 years will be eligible to participate in a pre-screening session to determine whether they meet inclusion criteria. During the pre-screening session, eligibility will be assessed with the Physical Activity Readiness Questionnaire for Everyone (2011) and the individual's blood pressure reading. Participants are eligible if they meet these criteria, complete the screening tools listed above, and do not meet any of the exclusion criteria listed below.

Exclusion Criteria:

* During the pre-screening session, eligibility will be assessed with the Physical Activity Readiness Questionnaire for Everyone (2011) and the individual's blood pressure reading. Individuals will not be eligible to participate if any of the following occur:

  1. The participant responds that they are or may be pregnant.
  2. The participant responds "Yes" to any question on the Physical Activity Readiness Questionnaire for Everyone with the exception of reporting a mental health condition (e.g., anxiety, depression, attention-deficit hyperactivity disorder) that is well controlled by medication and/or other therapies.
  3. The participant's blood pressure is 160 mm Hg or higher systolic or 90 mm Hg or higher diastolic.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Minutes spent engaging in physical activity during each phase | Participants are in the lab for one 1-hour session. These observational data will be recorded continuously (every second) during the 1-Hour session.
  Trained research assistants will use software to score time-stamped duration of engagement in physical activity (defined as walking or running on the treadmill).
Minutes spent engaging in sedentary activity during each phase | Participants are in the lab for one 1-hour session. These observational data will be recorded continuously (every second) during the 1-Hour session.
  Trained research assistants will use software to score time-stamped duration of engagement in sedentary activity (defined as sitting or standing).
Average heart rate for each phase | Participants are in the lab for one 1-hour session. The polar heart rate monitor will be worn at all times during the session and the device samples heart rate at least one time per second during the 1-Hour session.
  The heart rate monitor will sample and record heart rate on a second-by-second basis. The average heart rate will be calculated for each phase.
Real-time record of heart rate | Participants are in the lab for one 1-hour session. The polar heart rate monitor will be worn at all times during the session and the device samples heart rate at least one time per second during the 1-Hour session.
  The heart rate monitor will sample and record heart rate on a second-by-second basis and produce a time-stamped record that can be graphed and analyzed as time-series data.

SECONDARY OUTCOMES:
Real-time record of activity zone | Participants are in the lab for one 1-hour session. The polar heart rate monitor will be worn at all times during the session and the device samples heart rate at least one time per second during the 1-Hour session.
  The heart rate monitor will produce a record of activity level based on heart rate data and will produce a time-stamped record that can be graphed and analyzed as time-series data. The software calculates activity zone based on percentage of maximum heart rate. There are 5 zones of activity.
Average number of minutes in each activity zone during each phase | Participants are in the lab for one 1-hour session. The polar heart rate monitor will be worn at all times during the session and the device samples heart rate at least one time per second during the 1-Hour session.
  The heart rate monitor will produce a record of activity level based on heart rate data and will produce a time-stamped record. The software calculates the activity zone based on the percentage of maximum heart rate. Average number of minutes spend in each zone will be calculated for each phase.
Systolic and Diastolic Blood Pressure reading | Screening session and during the 1-hour session.
  Systolic or Diastolic Blood Pressure will be measured using a blood pressure monitor.
Duration of time spend engaging in each activity type. | Participants are in the lab for one 1-hour session. These observational data will be recorded continuously (every second) during the 1-Hour session.
  Trained research assistants will use software to score time-stamped duration of engagement. There will be 10 activity codes (Treadmill; Moving, Treadmill; Not Moving, Sitting, Standing, Watching screen (phone, computer, etc), Looking at paper or book, Sleeping or eyes closed, Other Leisure, Other gross-motor movement, and interacting with experimenter).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn M Kestner, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Observational & behavioral data collected during the proposed project will be made available (the tentative plan is to do so through The Research Repository @ WVU). Submitted data will conform with relevant data and terminology standards. All identifiable information will be removed to protect confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication for at least 5 years.
Access Criteria: Anyone interested in accessing the data.
URL: https://researchrepository.wvu.edu/